CLINICAL TRIAL: NCT06652607
Title: Evaluation of Biochemical Response as Prognostic Factor in Metastatic Castration-Sensitive Prostate Cancer and Analysis of Baseline Characteristics Between Patients With or Without PSA Value of 0.2 ng/dl.
Brief Title: PSA Biochemical Response as Prognostic Factor in Metastatic Castration-Sensitive Prostate Cancer
Acronym: PSA-DEEP02
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7039
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer; Metastatic Cancer; Castrate Sensitive Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — enzalutamide; apalutamide; darolutamide; Docetaxel; Abiraterone Acetate; Prednisone; Prednisolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Enzalutamide — The objective of the study is to assess survival in patients treated with Enzalutamide according to PSA response and to describe the baseline characteristics of patients with and without an optimal PSA response.
Drug: Apalutamide (Erleada™) 60 mg or 240 mg tablets — The objective of the study is to assess survival in patients treated with Apalutamide according to PSA response and to describe the baseline characteristics of patients with and without an optimal PSA response.
Drug: Darolutamide (Nubeqa®) 300 mg tablets — The objective of the study is to assess survival in patients treated with Darolutamide according to PSA response and to describe the baseline characteristics of patients with and without an optimal PSA response.
Drug: Taxotere (docetaxel) — The objective of the study is to assess survival in patients treated with Taxotere according to PSA response and to describe the baseline characteristics of patients with and without an optimal PSA response.
Drug: Abiraterone acetate + Prednisone or Prednisolone — The objective of the study is to assess survival in patients treated with Abiraterone according to PSA response and to describe the baseline characteristics of patients with and without an optimal PSA response.

SUMMARY:
Prostate cancer remains the most common malignancy in men in Europe. Over the last two decades, the treatment landscape for both localized and metastatic prostate cancer has been revolutionized. For patients with metastatic castration-sensitive prostate cancer (mCSPC), the primary treatment objectives are to delay progression to metastatic castration-resistant prostate cancer (mCRPC) and to improve overall survival (OS). Although patients with PC may initially respond to androgen deprivation therapy (ADT), progression to castration resistance occurs in 10-20% of patients within 5 years.

Primary ADT has been the standard of care for over 50 years. However, recent advancements have shifted treatment from ADT monotherapy for all mHSPC/mCRPC patients to more intensive approaches, which include combinations of ADT with new androgen receptor pathway inhibitors (ARPIs), chemotherapy, or both, tailored to tumor characteristics such as metastatic burden.

In clinical practice, a reduction in prostatic specific antigen (PSA) levels from baseline is commonly used to monitor disease control, particularly in the castration sensitive phase (both early and metastatic). For patients with mCSPC, a decrease in PSA levels signifies that the treatment is effective. Moreover, the depth, time and duration of this PSA reduction are linked to better clinical outcomes, including OS. Although more patients achieved an optimal PSA response with intensified ADT (with ARPI or docetaxel), those with a suboptimal response have a significantly worse survival rate. Several key studies have demonstrated that achieving undetectable PSA (≤0.2 ng/mL) is associated with better OS, irrespective of subgroups.

This study aims to evaluate patient survival based on PSA response and to describe baseline characteristics among patients with or without PSA response. Specifically, patients will be divided into two groups based on the achievement of PSA values ≤ 0.2 ng/dl, and overall survival (OS) and progression free survival (PFS) for each group will be evaluated. Clinical and laboratory information at baseline will be compared between the two groups. Baseline characteristics considered are histology, Gleason score, stage of disease, presence of genetic alterations, PSA values, sites and number of metastases, de novo or metachronous disease, high/low risk disease, high/low volume disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old;
* Men with histologically or cytologically confirmed adenocarcinoma of the prostate with evidence of metastases;
* ECOG performance status ≤2;
* Staging of disease with TC + bone scintigraphy or with PET PSMA/choline;
* Availability of baseline PSA and after six months (±1) from the beginning of the ADT;
* Ongoing or completed treatment with at least one ARPI among abiraterone acetate, apalutamide, darolutamide and enzalutamide;
* Adequate information about baseline demographic, biological, clinical and laboratory data;
* Signed informed consent form, or declaration in lieu of informed consent form, if applicable.

Exclusion Criteria:

* Patients without evidence of histological diagnosis of prostate cancer;
* No follow up visit after the beginning of therapy;
* No availability of baseline informations.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by metastatic castration sensitive prostate cancer who received the diagnosis from July 2022 treaded, and started androgen deprivation therapy plus one ARPI-based therapy.
Sampling Method: Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the survival based on the PSA response at six months from the beginning of ARPI in patients with mCSPC. | 4 years
  To evaluate the overall survival (OS) between patients with or without a PSA response ≤0.2 ng/ml at six months (from the beginning of ADT) in patients with mCSPC.

SECONDARY OUTCOMES:
To evaluate the efficacy of ARPI-based therapy based on the PSA response at six months from the beginning of ARPI in patients with mCSPC. | 4 years
  To evaluate the progression-free survival (PFS) between patients with or without a PSA response ≤0.2 ng/ml at six months (from the beginning of ADT).
To describe the baseline characteristics between patients with or without PSA response. | 4 years
  To describe the baseline clinical and biological characteristics between patients who achieved a PSA response ≤0.2 ng/ml at six months (from the beginning of ADT).
To describe the timing of PSA response | 4 years
  To describe the timing from the beginning of the ADT and the value ≤0.2 ng/dl among the responder patients.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Iacovelli, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC ONCOLOGIA MEDICA, Rome, Lazio, Italy